CLINICAL TRIAL: NCT01654484
Title: A Phase I/II, Randomized, Observer-masked, Placebo-and Active-controlled, Parallel-group, Multi-center Study Assessing the Safety and Efficacy of DE-117 Ophthalmic Solution in Subjects With Primary Open-angle Glaucoma or Ocular Hypertension
Brief Title: A Study Assessing the Safety and Efficacy of DE-117 Ophthalmic Solution in Patients With POAG or OHT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33-001
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — tafluprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Low Dose DE-117 (Experimental): Monotherapy
  Interventions: Drug: DE-117
- Medium Dose DE-117 (Experimental): Monotherapy
  Interventions: Drug: DE-117
- High Dose DE-117 (Experimental): Monotherapy
  Interventions: Drug: DE-117
- Low Dose DE-117 and 0.0015% tafluprost (Experimental): Adjunctive Therapy
  Interventions: Drug: DE-117 and 0.0015% tafluprost
- Med. Dose DE-117 and 0.0015% tafluprost (Experimental): Adjunctive Therapy
  Interventions: Drug: DE-117 and 0.0015% tafluprost
- High Dose DE-117 and 0.0015% tafluprost (Experimental): Adjunctive Therapy
  Interventions: Drug: DE-117 and 0.0015% tafluprost
- 0.0015% tafluprost (Active Comparator): Monotherapy
  Interventions: Drug: 0.0015% tafluprost
- Placebo (Placebo Comparator): Monotherapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DE-117 — Ophthalmic Solution, QD, 28 Days
  Arms: High Dose DE-117; Low Dose DE-117; Medium Dose DE-117
Drug: 0.0015% tafluprost — Ophthalmic Solution, QD, 28 days
  Arms: 0.0015% tafluprost
Drug: DE-117 and 0.0015% tafluprost — Ophthalmic Solutions, QD, 28 days
  Arms: High Dose DE-117 and 0.0015% tafluprost; Low Dose DE-117 and 0.0015% tafluprost; Med. Dose DE-117 and 0.0015% tafluprost
Drug: Placebo — Ophthalmic Solution, QD, 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of up to three concentrations of DE-117 ophthalmic solution (Low Dose, Medium Dose, and High Dose) as monotherapy and as adjunctive therapy (DE-117 ophthalmic solution with 0.0015% tafluprost) in subjects with primary open-angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
This is a two stage study.

Stage One will explore the dose response of three concentrations of DE-117 as monotherapy compared with 0.0015% tafluprost and placebo. The safety and efficacy of DE-117 as adjunctive therapy (with 0.0015% tafluprost) compared with 0.0015% tafluprost and placebo will also be evaluated. In addition, the additive effect of adjunctive therapy of each concentration will be compared with the corresponding monotherapy concentration.

Stage Two will assess the safety and efficacy of the optimal DE-117 concentration as monotherapy compared with 0.0015% tafluprost. The safety and efficacy of the optimal DE-117 concentration as adjunctive therapy (with 0.0015% tafluprost) compared with DE-117 monotherapy and 0.0015% tafluprost will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older
2. Current diagnosis of primary open-angle glaucoma or ocular hypertension in both eyes
3. Qualifying intraocular pressure (IOP) in at least one eye at Baseline

Exclusion Criteria:

1. Closed/barely open anterior chamber angle or a history of acute angle closure in either eye
2. Anticipate the need to initiate or modify medication (systemic or topical) that is known to affect intraocular pressure (IOP) during the study period
3. Females who are pregnant, nursing or planning a pregnancy
4. Presence of any abnormality or significant illness that could be expected to interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in intraocular pressure (IOP) on Day 29 at each scheduled time point | Day 28 T0 (08:00 ±30 mins), T0+2 hrs, T0+4 hrs, T0+8 hrs

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Santen Investigational Site, Newport Beach, California
  - Santen Investigational Site, Deerfield Beach, Florida
  - Santen Investigational Site, Largo, Florida
  - Santen Investigational Site, Morrow, Georgia
  - Santen Investigational Site, Roswell, Georgia
  - Santen Investigational Site, Rochester, New York
  - Santen Investigational Site, Cleveland, Ohio
  - Santen Investigational Site, Austin, Texas
  - Santen Investigational Site, Fort Worth, Texas
  - Santen Investigational Site, San Antonio, Texas